CLINICAL TRIAL: NCT02496689
Title: An Open-label, Multicenter, Expanded Access Program for Asfotase Alfa (Human Recombinant Tissue-nonspecific Alkaline Phosphatase Fusion Protein) Treatment for Patients With Infantile- or Juvenile-onset Hypophosphatasia (HPP)
Brief Title: Expanded Access Program for Asfotase Alfa Treatment for Patients With Infantile- or Juvenile-onset Hypophosphatasia (HPP)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AA-HPP-405
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia
Keywords: HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

INTERVENTIONS:
Biological: asfotase alfa — Patients participating in this program will receive 6 mg/kg/week asfotase alfa (administered at a dosage regimen of 1 mg/kg 6 times per week or 2 mg/kg 3 times per week at the discretion of the Investigator) by SC injection. During follow-up visits, dose adjustments to account for changes in body weight will be made. Additional incremental dose adjustments for lack of efficacy or safety reasons may also be decided upon by the Investigator in consultation with the Alexion Medical Monitor.

SUMMARY:
This clinical trial is being conducted in Hypophosphatasia, a bone disorder caused by gene mutation(s) resulting in bone defects. These gene mutations cause low levels of an enzyme needed to harden bone. The purpose of this study is to provide access to treatment in a disease where no approved treatment exists. This is an experimental treatment provided under specific treatment guidelines in which safety endpoints will be collected.

DETAILED DESCRIPTION:
U.S. sites participating in the expanded access program are closed to enrollment.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria for participation in this program:

1. Patient or parent (or legal guardian) must provide written informed consent prior to the performance of any program-related procedures and must be willing to comply with program procedures. Where appropriate and required by local regulations, patient assent for participation must also be obtained.
2. Patient must have a documented diagnosis of HPP as indicated by a documented history of HPP-related skeletal abnormalities and one or more of the following:

   * Documented tissue-nonspecific alkaline phosphatase (TNSALP) gene mutation(s)
   * Serum alkaline phosphatase (ALP) level below the age-adjusted normal range AND plasma pyridoxal-5'-phosphate (PLP) above the upper limit of normal at Screening. NOTE: Historical results for PLP may be used to determine patient eligibility. The criterion for plasma PLP is not applicable if the patient is receiving pyridoxine treatment.
3. Patient must have infantile- or juvenile-onset HPP, defined as documented onset of signs/symptoms of HPP prior to 18 years of age.
4. Male patient is:

   * Prepubertal; OR
   * Surgically sterile (defined as vasectomized for ≥6 months at Baseline); OR
   * Non-surgically sterile (defined as non-vasectomized or vasectomized for <6 months at Baseline) and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of two forms of birth control (at least one of which must be a barrier method) as described below starting at Baseline and continuing for 3 months after program completion.

     * Simultaneous use of condom, and for the female partner established use of hormonal contraceptives (eg, oral, injected, implanted) or intra-uterine contraceptive device
     * Simultaneous use of condom, and for the female partner occlusive cap (diaphragm or cervical/vault caps) with intravaginally applied spermicide
5. Female patient is:

   * Of non-childbearing potential, defined as:

     * Prepubertal; OR
     * Post-menopausal (defined as absence of menses for 12 months prior to Baseline or bilateral oophorectomy or hysterectomy with bilateral oophorectomy at least 6 months prior to Baseline); OR
     * Surgically sterile (defined as having hysterectomy or tubal ligation at least 6 months prior to Baseline) OR
   * Of childbearing potential, and:

     * Not sexually active; OR
     * Sexually active with non-sterile male spouse/partner (sterile male spouse/partner defined as a man vasectomized for ≥6 months) and must be using highly effective contraception consisting of two forms of birth control (at least one of which must be a barrier method) as described below and continuing for 3 months after program completion.
     * Simultaneous use of hormonal contraceptives (eg, oral, injected, implanted) or intra-uterine contraceptive device since at least 4 weeks prior to Baseline, and condom for the male partner
     * Simultaneous use of occlusive cap (diaphragm or cervical/vault caps) with intravaginally applied spermicide, and a condom for the male partner, since at least 14 days prior to Baseline
6. Male patients who are pubertal or post-pubertal and not surgically sterile (surgically sterile defined as vasectomized for ≥6 months) must agree to not donate sperm during program participation and for 3 months after program completion.
7. Female patients of childbearing potential (ie, those who are not prepubertal or postmenopausal or surgically sterile as defined in inclusion criteria 5 above) must have a negative urine or serum pregnancy test at Screening.

Exclusion Criteria

Patients will be excluded from participation in this program if they meet one or more of the following exclusion criteria:

1. Patient has geographic access to and qualifies for enrollment (as determined by the Sponsor and Investigator) in any other Alexion-sponsored clinical trials of asfotase alfa that are open to enrollment (eg, ENB-010-10).
2. Patient is pregnant, trying to become pregnant, or is lactating.
3. Patient has a documented sensitivity to any of the components of asfotase alfa.
4. Patient has serum calcium and/or phosphorus levels below the normal range at Screening.
5. Patient is currently enrolled in any other program or study involving an investigational new drug, device, or treatment for HPP (eg, bone marrow transplantation).
6. Patient has any other medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with program compliance, including all evaluations and follow-up activities. Patients who previously received treatment with asfotase alfa may be considered for enrollment.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Denker, MD, PhD, Study Director — Medical Monitor
Locations (5):
- United States (2):
  - Colorado Center for Bone Research, Lakewood, Colorado
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- France (3):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital des Enfants, Toulouse